CLINICAL TRIAL: NCT02842983
Title: Pilot Study: Echocardiographic and Hemodynamic Effects of Esmolol in Septic Shock Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: esmolol sepsis
Record Dates: First submitted 2016-07-14; First posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Shock, Septic
Keywords: Esmolol; Hypotension; Shock, Septic; Sepsis; Systemic Inflammatory Response Syndrome; Adrenergic beta-1 Receptor Antagonists; Adrenergic Antagonists; Pharmacologic Actions; Physiological Effects of Drugs
MeSH Terms: conditions — Shock, Septic; Hypotension; Sepsis; Systemic Inflammatory Response Syndrome | interventions — esmolol; Adrenergic beta-Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Esmolol (Experimental): After, at least six hours of hemodynamic optimization, patients with a hyperdynamic shock received a conventional management with a continuous infusion of Esmolol titrated to gain a 10% reduction in heart rate. This infusion is maintained for 72 hours.
  Interventions: Drug: Esmolol
- Control (No Intervention): Patients received conventional management of septic shock

INTERVENTIONS:
Drug: Esmolol — conventional management plus esmolol infusion
  Other Names: beta blockers
  Arms: Esmolol

SUMMARY:
After initial hemodynamic stabilization, 36 septic shock patients with heart rate > of 90 bpm and requiring norepinephrine to maintain mean arterial pressure (MAP) more than 65 mmHg will be randomised into two groups, esmolol group and control group. Patients allocated to esmolol group will receive a continuous esmolol infusion to maintain a lowering of heart rate of 10%. Norepinephrine will be titrated to achieve a MAP more than 65 mmHg. To investigate myocardial performance, the investigators will assess Tissue Doppler imaging by echocardiography and hemodynamic measures. Data will be obtained at baseline ,after esmolol infusion once achieved the predefined heart rate threshold and 72hours after esmolol infusion.

DETAILED DESCRIPTION:
primary outcome were determined according to our previous study of tissue doppler.

ELIGIBILITY:
Inclusion Criteria:

* septic shock
* fluid optimization
* with a cardiac index > 3 l/min/m2
* Heart Rate >90 /min

Exclusion Criteria:

* Cardiogenic shock
* Bradycardia
* History of Severe Asthma
* Indications against Esmolol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Echocardiographic assessment of heart function | over a period of 72 hrs
  peak systolic velocity measured at the mitral annulus decreased 30% compared with control group

SECONDARY OUTCOMES:
Effects on vasopressor requirement | over a period of 72 hrs
  Dosage of norepinephrine increased 100% compared with control group
90-day hospital mortality | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Yong-tai Liu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to share individual participant data.